CLINICAL TRIAL: NCT04951596
Title: Application Value of Precision Management Standard of Bone Marrow Infusion in Acute and Critical Patients
Brief Title: Management Standard of Bone Marrow Infusion in Acute and Critical Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-170
Record Dates: First submitted 2021-06-17; First posted 2021-07-07 (Actual); Last update posted 2021-07-07 (Actual); Status verified 2021-01

CONDITIONS: Emergency Patients
Keywords: Acute and critically ill patients; Intraosseous infusion; Management standards

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Investigate the current situation — Investigate the current situation of infusion treatment for acute and critical patients in 2 hospitals in the province

SUMMARY:
As the spike in the number and severity of patients with critical patients, then quickly effective transfusion treatment demand becomes more and more serious, and the pattern of infusion pathways have traditionally used already can not adapt to this change, therefore, an urgent need to establish a set of is in line with international standards and accord with the situation of our country is simple, effective and scientific accuracy of IO management solution. In order to ensure the safety of the treatment of acute and critical patients, and in the province and even domestic experts recognized and promoted the application.

DETAILED DESCRIPTION:
1. Investigate the current situation of infusion treatment for critical and critical patients in two hospitals in the province, the cognition of medical staff in critical and critical units on IO, IO training and assessment, and continuous quality improvement, etc. A comprehensive understanding of the needs of medical staff in the acute critical care unit for the refined IO management standard, including the analysis of the application of the standard in some hospitals.
2. Clarify and refine the contents of relevant indexes of IO management standards to form a standardized, scientific, unified and simple way to quickly judge difficult vessels. Defining the appropriate infusion access, infusion tool, puncture site, infusion speed, infusion effect, patient outcome, complications, indications, contraindication, infusion risk management, relevant personnel training and assessment, and continuous quality improvement as indexes.
3. On the basis of the standards of existing guidelines, a reasonable observation time range and the number of puncture times consistent with the first infusion puncture were established.

ELIGIBILITY:
Inclusion Criteria:

* 1.Emergency medical staffMore than two years of critical work experience 2.Volunteer to participate in research

Exclusion Criteria:

* Patients who have neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Emergency medical staff
  2. Bone marrow cavity catheterization patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
complications in patients with intraosseous infusion | one and a half years
  The number of complications occurred in the bone marrow cavity was calculated
time of infufusion access establishment for patients | one and a half years
  The time of catheterization for each bone marrow cavity puncture was recorded
Success rate of infusion access establishment | one and a half years
  The success rate of establishing the infusion access was calculated

CONTACTS AND LOCATIONS:
Overall Officials: minfei yang, Principal Investigator — 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China
Locations (2):
- China (2):
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hangzhou, Zhejiang
  - 2nd Affiliated Hospital, School of Medicine, Zhejiang University, China, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Voigt J, Waltzman M, Lottenberg L. Intraosseous vascular access for in-hospital emergency use: a systematic clinical review of the literature and analysis. Pediatr Emerg Care. 2012 Feb;28(2):185-99. doi: 10.1097/PEC.0b013e3182449edc. PMID 22307192
- [Result] Wampler D, Schwartz D, Shumaker J, Bolleter S, Beckett R, Manifold C. Paramedics successfully perform humeral EZ-IO intraosseous access in adult out-of-hospital cardiac arrest patients. Am J Emerg Med. 2012 Sep;30(7):1095-9. doi: 10.1016/j.ajem.2011.07.010. Epub 2011 Oct 24. PMID 22030185
- [Result] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Result] Whitney R, Langhan M. Vascular Access in Pediatric Patients in the Emergency Department: Types of Access, Indications, and Complications. Pediatr Emerg Med Pract. 2017 Jun;14(6):1-20. PMID 28562239